CLINICAL TRIAL: NCT02700646
Title: Improving Motor Skill Development in Infants After Cardiac Surgery
Acronym: DAISY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Karen Uzark, Professor of Cardiac Surgery and Associate Professor of Pediatric Cardiology, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HUM00107611
Record Dates: First submitted 2016-03-02; First posted 2016-03-07 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard care (No Intervention): Standard care comparison
- inpatient (Experimental): Inpatient recommendations to parents regarding infant motor activities
  Interventions: Behavioral: Developmental recommendations; Behavioral: Standard care
- inpatient/outpatient (Experimental): Inpatient and outpatient recommendations to parents regarding infant motor activities
  Interventions: Behavioral: Developmental recommendations; Behavioral: Standard care

INTERVENTIONS:
Behavioral: Developmental recommendations
  Arms: inpatient; inpatient/outpatient
Behavioral: Standard care — standard care
  Arms: inpatient; inpatient/outpatient

SUMMARY:
The purpose of this study is to learn more about developmental behaviors and to examine changes in developmental progress related to motor activities among a group of infants who received open heart surgery within the first three months of life.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) and the need for life-saving heart surgery and intensive care during infancy may have effects on infant behavior and development. Children who require open heart surgery before their first birthday are vulnerable to developmental delays, especially related to motor skills (mobility) in the first year of life. Early delays in gross motor functioning (e.g., rolling, crawling, walking) have implications for learning and psychosocial development through adulthood. To date, no interventions to improve the gross motor functioning of children born with CHD have been developed. The purpose of this study is to learn more about developmental behaviors and to examine changes in developmental progress related to motor activities among a group of infants who received open heart surgery within the first three months of life. Activities will be tailored based on the individual infant's motor ability and medical status.

ELIGIBILITY:
Inclusion Criteria:

* All hospitalized infants under age 4 months having cardiac surgery before age 3 months
* Intubation >/= 24 hours </= 14 days

Exclusion Criteria:

* Prematurity </= 36 weeks gestation
* Pre-operative clinical evidence of a central nervous system (CNS) anomaly or history of CNS insult

Max Age: 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Gross Motor Scale score | 3 months after hospital discharge
  Alberta Infant Motor Scale (AIMS) score

CONTACTS AND LOCATIONS:
Overall Officials: Karen Uzark, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States